CLINICAL TRIAL: NCT07366255
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Evaluate the Safety and Efficacy of Tripalmitoleoylglycerol for the Treatment of Dermatitis.
Brief Title: Safety and Efficacy of Tripalmitoleoylglycerol in Dermatitis: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LL-KY-2025270-02; 82372532, 82202468 (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2026-01-17; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Skin Barrier to Water Loss; PASI /SCORAD Index

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Sedentary + Placebo (Placebo Comparator): * Population/behavior: Sedentary (no regular exercise habit, <600MET-min/week)
  * Topical treatment: Placebo topical formulation
  * Duration: 7 days (topical once daily)
  Interventions: Other: Placebo topical intervention
- Arm 2: Sedentary + Tripalmitoleoylglycerol (Experimental): * Population/behavior: Sedentary (no regular exercise habit, <600MET-min/week)
  * Topical treatment: 0.5% Tripalmitoleoylglycerol topical formulation
  * Duration: 7 days (topical once daily)
  Interventions: Other: 0.5% Tripalmitoleoylglycerol topical intervention
- Arm 3: Exercise + Placebo (Experimental): * Population/behavior: Regular aerobic exercise habit, , >600MET-min/week, <3000MET-min/week
  * Topical treatment: Placebo topical formulation
  * Duration: 7 days (topical once daily)
  Interventions: Other: Placebo topical intervention
- Arm 4: Exercise + Tripalmitoleoylglycerol (Experimental): * Population/behavior: Regular aerobic exercise habit, , >600MET-min/week, <3000MET-min/week
  * Topical treatment: 0.5% Tripalmitoleoylglycerol topical formulation
  * Duration: 7 days (topical once daily)
  Interventions: Other: 0.5% Tripalmitoleoylglycerol topical intervention

INTERVENTIONS:
Other: Placebo topical intervention — Placebo topical intervention applied continuously for 7 days (once daily).
  Arms: Arm 1: Sedentary + Placebo; Arm 3: Exercise + Placebo
Other: 0.5% Tripalmitoleoylglycerol topical intervention — 0.5% Tripalmitoleoylglycerol topical intervention applied continuously for 7 days (once daily).
  Arms: Arm 2: Sedentary + Tripalmitoleoylglycerol; Arm 4: Exercise + Tripalmitoleoylglycerol

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial is designed to evaluate the safety and efficacy of topical palmitoleic acid glyceride supplementation in improving skin barrier impairment associated with chronic dermatitis, with a particular focus on the interaction between physical activity, skin microbiota, and lipid metabolism.

Emerging evidence suggests that regular physical activity reshapes the skin microenvironment, including alterations in sebaceous lipid composition and enrichment of Staphylococcus epidermidis, which possesses lipase activity capable of metabolizing glycerides into bioactive fatty acids. Palmitoleic acid, a key lipid metabolite derived from palmitoleic acid glycerides, has demonstrated anti-inflammatory and barrier-protective properties in preclinical and clinical settings. However, it remains unclear whether restoring exercise-associated lipid metabolites through topical application can improve skin barrier dysfunction in individuals with chronic dermatitis, and whether physical activity status modifies therapeutic efficacy.

Research Objectives：

1. Does topical application of low-concentration palmitoleic acid glyceride improve skin barrier function, as measured by transepidermal water loss (TEWL), in individuals with chronic dermatitis?
2. Does physical activity status influence the therapeutic response to palmitoleic acid glyceride treatment?
3. Are improvements in skin barrier function associated with changes in skin microbiota composition, microbial lipase activity, and lipid metabolism at the skin surface?

Study Design and Group Allocation：

Eligible male participants aged 18-59 years with clinical manifestations of chronic dermatitis and evidence of skin barrier impairment will be enrolled. Based on physical activity levels defined according to World Health Organization guidelines, participants will be stratified into physically inactive/insufficiently active and physically active/highly active groups. Within each stratum, participants will be randomly assigned in a 1:1 ratio to receive either topical palmitoleic acid glyceride or placebo, resulting in four study groups:

1. Inactive Placebo Group: No regular physical activity; topical placebo.
2. Inactive Intervention Group: No regular physical activity; topical palmitoleic acid glyceride.
3. Active Placebo Group: Regular moderate-intensity aerobic activity; topical placebo.
4. Active Intervention Group: Regular moderate-intensity aerobic activity; topical palmitoleic acid glyceride.

Participant Procedures：

1. Daily topical application of either 0.5% palmitoleic acid glyceride or placebo to a predefined skin lesion area for 7 consecutive days.
2. Non-invasive assessment of skin barrier function, including TEWL measurements, at baseline and after completion of the intervention.
3. Clinical evaluation of skin symptoms, including erythema, scaling, and pruritus, using standardized scoring systems (PASI or SCORAD, as appropriate).
4. Collection of skin swab samples for microbiome and metabolomic analyses to assess microbial lipase activity and palmitoleic acid production.
5. A subset of participants will undergo skin biopsy for histological and immunohistochemical analyses.
6. Weekly follow-up assessments to monitor treatment adherence and record any adverse events, particularly local skin reactions.

This study seeks to elucidate a novel exercise-microbiota-lipid axis in skin barrier regulation and to provide translational evidence for metabolite-based therapeutic strategies in chronic inflammatory skin diseases.

ELIGIBILITY:
Inclusion Criteria：

1. Participants must meet the latest physical activity guidelines issued by the World Health Organization and the U.S. Department of Health and Human Services, defined as follows:

   Inactive: No moderate- or vigorous-intensity physical activity beyond activities of daily living; Insufficiently active: Less than 150 minutes of moderate-intensity physical activity per week or less than 75 minutes of vigorous-intensity physical activity per week; Active: Approximately 150-300 minutes of moderate-intensity physical activity per week; Highly active: More than 300 minutes of moderate-intensity physical activity per week.

   Participants classified as inactive or insufficiently active will be assigned to the control group, whereas those classified as active or highly active will be assigned to the exercise group.
2. Presence of clinical manifestations of skin barrier impairment, such as skin dryness, erythema, scaling, or pruritus;
3. Voluntary participation with full understanding of the study and provision of written informed consent;
4. Age between 18 and 59 years, with generally good health status;
5. No use of any medications or probiotic treatments within the past 6 months;
6. No diagnosed skin diseases or skin injuries.

Exclusion Criteria：

1. History of allergy or known hypersensitivity to probiotics, placebo, or investigational products;
2. Presence of active skin diseases or other severe systemic diseases;
3. Pregnant or breastfeeding women;
4. Use of medications that may affect skin barrier function, such as corticosteroids or immunosuppressive agents;
5. Any other condition deemed inappropriate for study participation by the investigators, including but not limited to participants considered unreliable or unable to understand or comply with study assessments

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-12-28 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-02-04 (Estimated)

PRIMARY OUTCOMES:
1. Mean change in transepidermal water loss (TEWL, g/h/m²) at the intervention site | Baseline (Day 0) through Day 7 after intervention
  Transepidermal water loss (TEWL) will be assessed on the marked lesion area using a Tewameter (TM300) under standardized environmental conditions (controlled temperature and humidity). At each assessment, TEWL will be measured at three predefined points within the intervention area, and the mean value will be calculated.
  The primary outcome is defined as the mean change in TEWL (g/h/m²) from baseline (Day 0) to Day 7 after intervention. Lower TEWL values indicate improved skin barrier function.
2. Change in clinical dermatitis severity assessed by PASI or SCORAD index | Baseline (Day 0) through Day 7 after intervention
  Description:
  Clinical severity of dermatitis will be evaluated in the intervention area by trained investigators using standardized scoring systems.
  Psoriasis patients will be assessed using the Psoriasis Area and Severity Index (PASI).
  Atopic dermatitis patients will be assessed using the SCORing Atopic Dermatitis (SCORAD) index.
  The outcome is defined as the change in PASI or SCORAD score from baseline (Day 0) to Day 7 after intervention, reflecting improvement in erythema, scaling, and pruritus.

SECONDARY OUTCOMES:
3. Skin surface lipase activity and palmitoleic acid production assessed by skin swab metabolomics | Baseline (Day 0) through Day 7 after intervention
  Skin swab samples will be collected from the intervention site in both sedentary and exercise groups at baseline and after intervention. Targeted metabolomic analyses will be performed to evaluate skin surface lipase activity and the metabolism of glycerides into palmitoleic acid.
  The outcome is defined as the change in skin surface lipase activity and palmitoleic acid levels between baseline and post-intervention.
4. Immunohistochemical analysis of skin biopsy samples | Day 7 after intervention
  Skin biopsy samples (3-4 mm) will be obtained from a subset of participants (3-4 individuals per group) in both sedentary and exercise groups. Immunohistochemical staining will be performed to assess changes in inflammatory markers and skin barrier-related proteins.
  This outcome is exploratory and intended to support mechanistic interpretation of clinical findings.

IPD SHARING:
Plan to Share IPD: No